CLINICAL TRIAL: NCT03452046
Title: Inferior Vena Cava Indexes (Collapsibility, Distensibility, Delta) in Positive Pressure Supports and Prediction Ability of Intravascular Volume Status in ICU Patients
Brief Title: Inferior Vena Cava Indexes in Positive Pressure Supports
Status: Completed | Type: Observational
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aykut Saritas, Principal Investigator, Tepecik Training and Research Hospital
Other Study IDs: Tepecik
Record Dates: First submitted 2018-02-25; First posted 2018-03-02 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Positive-Pressure Respirations; Respiratory Failure
Keywords: Ultrasound,inferior vena cava, positive pressure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Central Venous Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PS 10 mmHg, PEEP 5 mmHg: IVC diametres, CI-IVC, distensibility and delta index measurements using by ultrasound. Central venous pressure correlation with IVC index
  Interventions: Other: IVC diametres
- PS 10 mmHg PEEP 0 mmHg: IVC diametres, CI-IVC, distensibility and delta index measurements using by ultrasound. Central venous pressure correlation with IVC index
  Interventions: Other: IVC diametres
- PS 0 mmHg PEEP 5 mmHg: IVC diametres, CI-IVC, distensibility and delta index measurements using by ultrasound. Central venous pressure correlation with IVC index
  Interventions: Other: IVC diametres
- t tube (PS 0 mmHg PEEP 0mmHg): IVC diametres, CI-IVC, distensibility and delta index measurements using by ultrasound. Central venous pressure correlation with IVC index
  Interventions: Other: IVC diametres

INTERVENTIONS:
Other: IVC diametres
  Other Names: Measurement of central venous pressure; Positive pressure supports

SUMMARY:
Collapsibility (CI-IVC), distensibility (dIVC) and delta (ΔIVC) indices, which are dynamic measures of inferior vena cava (IVC) diameter, are used to assess the intravascular volume status in critically ill patients. Positive pressure support (PS) has been shown to induce IVC diameter distention by increasing intrathoracic pressure, and high positive expiratory pressure (PEEP) decreases the CI-IVC percentage (4). During Triggered positive pressure support it is necessary to clarify which IVC index is valid for measuring the volume status.it is aimed to compare the IVC indexes (CI-IVC, DIVC, ΔIVC), positive rate of change with pressure, correlation with central venous pressure and accurate prediction of volume status in patients with different positive pressure support.

DETAILED DESCRIPTION:
The IVC diameters at different pressure supports were measured by the same clinician after obtaining a clear image of where the US and IVC measurements were made and the probe stabilization was achieved. He performed the procedure of changing the pressure supports, a blind independent intensive care physician without working, and recorded the applied pressure supports respectively. The different pressure supports applied are as follows:

1. PS 10 mmHg-PEEP 5 mmHg,
2. PS 0 mmHg- PEEP 5 mmHg
3. PS 10 mmHg- PEEP 0 mmHg.
4. T-tube (PS 0 mmHg-PEEP 0 mmHg)

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Current use of mechanical ventilation through an endotracheal tube.

Exclusion Criteria:

* Profound Hypoxia defined as a fraction of inspired oxygen requirement >90% or a PEEP >10 mmHg
* Patient-ventilator desynchrony or active agitation
* Unstable O2 requirement
* Cardiovascular instability
* Current PEEP requirements of >10 mmHg
* Current oxygen saturation (SpO2) of <88%.
* High intra abdominal pressure
* Right cardiac failure
* Morbid obesity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatient sample
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Determine the effect of positive pressure on IVC collapsibility index | 12 month
  Determine the effect on CI-IVC of an increase in positive end-expiratory pressure and pressure support
Determine the effect of positive pressure on IVC distensibility index | 12 month
  Determine the effect on distensibility index of an increase in positive end-expiratory pressure and pressure support
Determine the effect of positive pressure on IVC delta index | 12 month
  Determine the effect on delta index of an increase in positive end-expiratory pressure and pressure support

SECONDARY OUTCOMES:
Determine the effect of positive pressure on central venous pressure | 12 month
  Determine the effect on central venous pressure of an increase in positive end-expiratory pressure and pressure support

CONTACTS AND LOCATIONS:
Overall Officials: Tepecik Training and Research Hospital, Principal Investigator — Tepecik Training and Research Hospital
Locations (1):
- Tepecik Research and Training Hospital, Izmir, Konak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided